CLINICAL TRIAL: NCT01625052
Title: Determination of the Optimal Approach to Select the Best Size of BASKA Mask to Use in Male Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, John Laffey, Professor of Anaesthesia and Critical care, Consultant Anaesthetist, University College Hospital Galway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.A.653
Record Dates: First submitted 2012-03-23; First posted 2012-06-21 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Determination of the Best Predictor for Correct Baska Mask Size
Keywords: mask size; Baska mask; supraglottic airway; airway management
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baska (Experimental)
  Interventions: Device: Placement and use of Baska mask

INTERVENTIONS:
Device: Placement and use of Baska mask — use of Baska mask as component of standard general anaesthetic

SUMMARY:
The investigators group has performed a number of studies on novel airway devices, including an observational study on the performance of a new supraglottic airway named Baska mask. In this new study the investigators wish to determine which criteria best predict the correct size of the Baska mask to be used in male patients

DETAILED DESCRIPTION:
Our observational study of the performance of the Baska mask suggests that this novel supraglottic airway has promise as an alternative to the current standard device, the laryngeal mask airway (LMA). Our results indicate that while the manufacturer weight criteria work reasonably well in females this may not be the case in males. The investigators wish to determine how well the manufacturer recommended sizing criteria for the Baska mask work in males.

This study is designed to determine which criteria best predict the correct size Baska mask to use in male patients. In addition the investigators will monitor the performance and safety of this device (insertion success rate, seal pressures, time to and ease of insertion, failure rate, complications etc)

ELIGIBILITY:
Inclusion Criteria:

* Male
* Written informed consent
* ASA 1-3
* No relevant allergies
* Body-mass index (BMI) 20-35
* Age 16-85
* Non-urgent surgery of planned duration 0.25-4 hrs

Exclusion Criteria:

* Inability of patient/parent to understand or consent for the trial
* Neck pathology
* Previous or anticipated problems with the upper airway or upper GI tract (reflux, hiatus hernia, oropharyngeal tumour, upper respiratory tract infection in the last 10 days)
* BMI > 35
* Predicted or previously documented difficult airway
* Increased risk for Gastric Aspiration
* Current participation in another Clinical Study

Ages: 16 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Determination of the best predictor for successful Baska mask size | From the moment of preoperative assessment until the moment of mask placement, an expected average of 3 hours.
  We will evaluate the correlation between certain patient characteristics (including, but not limited, to actual and ideal body weight; height) and the size of the Baska mask used successfully in each patient.

SECONDARY OUTCOMES:
insertion success rate of the device | within 30 min of anaesthesia commencement
device airway leak pressure | within 30 min of anaesthesia commencement
device insertion time | within 30 min of anaesthesia commencement
  the time from the moment the device is touched until successful ventilation is achieved or device is removed.
ease of insertion of device | within 30 min of anaesthesia commencement
  we will use 10cm visual analogue scale
complications | from the moment anaesthesia commenced up to the first postoperative day, an expected average of 30 hours.
  Complications during insertion, maintenance and removal and in the postoperative period (in PACU and next day follow up) List of complications (not exhaustive): desaturation episodes, loss of airway with need to manipulate mask/switch to alternative device, lip/teeth damage, regurgitation, aspiration, laryngospasm, blood staining on mask removal)
Patient comfort | from the moment patient awake up to third postoperative day, an expected average of 80 hours.
  We will record throat pain, dysphonia and dysphagia using 10 point verbal rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: John G Laffey, FFARCSI, Principal Investigator — National University of Ireland, Galway, and Galway University Hospitals
Locations (1):
- Galway University Hospitals, Galway, Galway, Ireland